CLINICAL TRIAL: NCT01169428
Title: Mindfulness Based Weight Loss Maintenance
Brief Title: Engaging Motivation for the Prevention of Weight Regain
Acronym: EMPOWER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Pennsylvania (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00013688; U01AT004159 (NIH)
Record Dates: First submitted 2010-07-22; First posted 2010-07-26 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Obesity
Keywords: Mindfulness-Based Weight Loss Maintenance; prevention of weight regain; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Behavioral Weight-Loss Maintenence (Active Comparator): Attention/Education/Support Control
  Group designed to control for educational content as well as multiple nonspecific treatment factors (e.g., support, time invested, leader attention, positive expectancy)
  Interventions: Behavioral: Behavioral: Standard Behavioral Weight-Loss Maintenence
- Behavioral: Mindfulness Based Weight Loss Maintenance (MBWLM) (Active Comparator): This mindfulness-meditation based intervention is designed to increase awareness of the factors that affect weight loss maintenance after successful weight loss.
  Interventions: Behavioral: Mindfulness Based Weight Loss Maintenance (MBWLM)

INTERVENTIONS:
Behavioral: Mindfulness Based Weight Loss Maintenance (MBWLM) — This mindfulness-meditation based intervention is designed to increase awareness of the factors that affect weight loss maintenance after successful weight loss. Mindfulness meditation is a technique for training awareness. The program will train subjects to increase awareness of the somatic, cognitive, affective, interpersonal and environmental factors that mediate eating and physical activity by incorporating empirically-supported and theoretically-synergized components, including: general mindfulness meditation skills, mindful and intuitive eating, appetite-satiety awareness, mindful movement and yoga, a mindful approach to exercise engagement, and training in enhancing emotion regulation and stress management skills. In addition, the MBWLM group will be supported by Maintenance Partners who are trained as Integrative Health Coaches.
  Arms: Behavioral: Mindfulness Based Weight Loss Maintenance (MBWLM)
Behavioral: Behavioral: Standard Behavioral Weight-Loss Maintenence — Attention/Education/Support Control group, designed to control for educational content as well as nonspecific treatment factors [e.g., natural history (time), amount of time and energy spent in the intervention, attention by group leaders, social support, as well as information & education]. Like the experimental group(MBWLM), this group meet once a week for 2 hours during the 12-week intervention, and then at 4 weeks, 8 weeks, and 12 weeks post the 12 week intervention. Participants also receive the same amount of telephonic support through Maintenance Partners as the experimental group, but their Maintenance Partners employed empathic listening only rather than myriad coaching techniques.
  Arms: Standard Behavioral Weight-Loss Maintenence

SUMMARY:
The purpose of this study is to determine whether a 12 week Mindfulness-Based Weight Loss Maintenance (MBWLM) intervention is effective in maintaining recent loss of 10% or more of initial body weight.

DETAILED DESCRIPTION:
Obesity is now recognized as the 2nd leading cause of preventable death in the U.S. and is associated with significant impairment. While structured behavioral regimes typically lead to significant weight loss, a burgeoning literature reveals less encouraging results for weight loss maintenance (WLM). Hence, innovative approaches to WLM are necessary to buffer against disease risks associated with weight regain. Interventions utilizing mindfulness meditation show promise in treating unhealthy eating behaviors and other obesity-related problems, including mood, blood sugar control and addiction. By enhancing self-awareness and emotion regulation, such interventions may be particularly useful in facilitating the internalization of healthy behavior change. The proposed study aims to develop a novel intervention to promote WLM. Specifically, we will develop a 12 week Mindfulness-Based Weight Loss Maintenance (MBWLM) intervention and test its efficacy against an attention/education/support control (ASC) condition in a two-arm RCT of overweight and obese (BMI > 25) men and women (N=95) who recently lost at least 10% of their initial body weight via non-surgical means. The primary endpoint will be percent change in weight from baseline to 12-month follow-up. We are also interested in testing the efficacy of the MBWLM program on improving secondary outcomes, including obesity/adiposity, health behaviors, and psychological well-being. In addition, we will study the impact of MBWLM on glucose metabolism, appetite/food intake regulation, and systemic inflammation. Outcome data will be collected at baseline, post-intervention, 6-month follow-up and 12-month follow-up. Multilevel ("mixed-effects") modeling will be used to test between-group differences on primary and secondary endpoints. Further, path analysis will be used to investigate mechanisms underlying successful WLM. Taken together, these data could provide support for the integration of mindfulness meditation into comprehensive treatment programs for obesity and weight management.

ELIGIBILITY:
Inclusion Criteria: 1) Gender: Men and women. 2) Ethnicity: Any, with over-sampling of African-Americans. 3) Age: >18 4) Weight: BMI > 20 at study entry. 5) Documented (by physician, community weight loss program, personal friend or family member) weight loss of at least 9% of total body weight completed within the previous 3 year period and not regained greater than half of the 9% loss.

6) Planning to be in the area through the length of follow-up. 7) Availability of telephone. 8) English-speaking and English-literate. 9) Commitment to attend all treatment and assessment appointments. 10) If on medication that may affect outcome variables, on stable dose with willingness to remain at that dose from baseline through end of weekly (12-week) intervention and 12 month follow-up, unless physician orders otherwise.

11) Willingness to not engage in any other formal weight loss program through the 12 month follow-up.

12) Provides Informed consent. 13) Participants can have a weight loss or gain of more than 8.8lbs within the 3 month period prior to enrollment. However, due to the possibility that this will influence baseline inflammatory bio markers we will document the amount of self-reported weight change within the 3 month period prior to their baseline lab appointment.

Exclusion Criteria:

1. Concurrent participation in a structured weight loss program, fad diet or use of weight loss medication or herbal supplements during 15 month course of the trial. If has been taking a weight loss medication or supplement, must go through a 1 month washout period before enrollment.
2. Previous weight reduction surgery, or initiating weight reduction surgery during the 15 month study period.
3. Inability to participate fully or behave appropriately in the group setting, as observed by (a). interviewing clinician and evidenced by two or more of the exclusionary criteria on the Appropriateness for Group Participation Behavioral Checklist or (b) baseline acknowledgement of substance abuse, psychotic episode(s), psychiatric hospitalization or history of self-harm within the past 2 years, or current suicidal or homicidal ideation.
4. Unstable medical condition, medical condition underlying weight or eating problems (e.g., Blood sugar greater than 350, Cancer and currently receiving radiation or chemo treatment, Cushing's Syndrome; thyroid disorder) or medical condition requiring strict dietary regimen.
5. Pregnant, breast-feeding, or unwilling to take contraceptive measures to prevent pregnancy during the 15 month study. If a woman has recently been pregnant, is currently nursing, or recently quit nursing, she must have stopped nursing and had 3 normal menstrual cycles or be using approved contraceptive measures for 3 months before being eligible.
6. Meeting diagnostic criteria for purging bulimia.
7. More than 1.5 hours of exposure to meditation-based eating or weight control techniques.
8. More than 60 minutes per week, for a consecutive 4 week time period, during the last 2 years, of regular sitting (Mindfulness Based Stress Reduction, Transcendental Meditation, or other meditation practice) meditation practice.
9. Not willing to be randomized.
10. No other household members can participate.
11. Baseline glucometer reading of >125 for previously unknown diabetics, as this is likely to indicate undiagnosed diabetes that would require more intensive treatment.
12. Known diabetes likely to require more intensive treatment, defined as a baseline glucometer reading > 350 or the inability to maintain a stable diabetes medication regimen for the previous 6 months.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2007-07; Primary Completion 2009-07 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Weight Loss Maintenance | 16-month
  Our primary endpoint will be an evaluation of differential weight loss maintenance (WLM) or weight regain between the two conditions. All weight measures will be taken on the Tanita scale in a standardized fashion, in the morning following a 12 hour fast, after voiding and in bare feet while wearing a standardized outfit.

SECONDARY OUTCOMES:
Body Mass Index | 16-month
  BMI is the most widely accepted indicator of overweight and obesity.
Waist circumference | 16 month
  Waist circumference will be assessed using methods prescribed by the United States Department of Health and Human Services. The point of measurement will be determined by locating the right iliac crest.
Percent Body Fat | 16 month
  Total body fat will be assessed using a bioelectrical impedance scale (Tanita Scale).
Psychological outcomes and lifestyle behavior | 16-month
  Questionnaires used to measure these outcomes, included POMS,PSS,SF-12, BES,IES,IPAQ,Modified Block Food Frequency Questionnaire,CAMS-R, 5-Factor Mindfulness Questionnaire,TAS-20
Biological markers of appetite | 16 months
  Assessed by serum Leptin, Ghrelin, PYY
Glucose metabolism | 16 months
  Evaluated by fasting serum glucose, postprandial glucose, fasting insulin, postprandial insulin, hemoglobin A1C
Biological markers of inflammation | 16 months
  Inflamation assessed by serum Interleukin-6 and serum C-Reactive Protein

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Q Wolever, PhD, Principal Investigator — Duke University; Michael Baime, M.D, Principal Investigator — University of PENN, Program for Stress Management
Locations (2):
- United States (2):
  - Duke University - Duke Integrative Medicine, Durham, North Carolina
  - University of Pennsylvania, Program for Mindfulness, Philadelphia, Pennsylvania